CLINICAL TRIAL: NCT04171492
Title: A Multicenter, Randomized Controlled Trial, Prospectively Evaluating the Clinical Utility of the Nodify XL2 Proteomic Classifier in Incidentally Discovered Low to Moderate Risk Lung Nodules
Brief Title: Nodify XL2 Classifier Clinical Utility Study in Low to Moderate Risk Lung Nodules
Acronym: ALTITUDE
Status: Active, not recruiting | Type: Observational
Sponsor: Biodesix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BDX-CD-003
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Nodule Solitary Pulmonary; Non-small Cell Carcinoma
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nodify XL2 plasma sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Open Label: Nodify XL2 results will be reported to the investigator and available to the subject.
- Blinded: Nodify XL2 results will not be available to the investigative site or subject.

SUMMARY:
This study evaluates the how addition of the Nodify XL2 test result impacts the clinical management of newly identified solid lung nodules assessed as low to moderate risk of cancer.

DETAILED DESCRIPTION:
A multicenter, randomized controlled study with a blinded control arm. Open label arm is observational for lung nodule management. The clinical trial will evaluate the clinical utility of the Nodify XL2 integrated classifier when used in the clinical management of newly identified solid lung nodules assessed as < 50% risk of cancer by Mayo risk prediction algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent to participate in the study and agrees to comply with all protocol requirements
2. Subject is > 40 years of age at the time of the discovery of the lung nodule of concern
3. Subject's lung nodule of concern meets the following:

   * Was incidentally identified or detected during lung cancer screening
   * Is a solid nodule
   * Has maximal dimension of > 8mm and < 30mm
4. The first CT scan identifying the lung nodule of concern was performed within 60 days of subject enrollment
5. The pre-test risk of cancer as determined by the Mayo risk prediction algorithm is 65% or less

Exclusion Criteria:

1. Nodule work-up at the time of subject enrollment indicating any prior attempted or completed diagnostic biopsy procedure or blood-based testing for the lung nodule of concern
2. Nodule of concern is part-solid or Ground Glass Opacity (GGO)
3. Prior diagnosis of lung cancer
4. Any active cancer within 5-years of nodule detection, with the exception of non-melanoma skin cancer
5. Administration of blood products (i.e. packed red blood cells, fresh frozen plasma, or platelets) within 30 days of subject enrollment
6. Concurrent participation in any unrelated clinical trial that may impact or alter the management of the subject's nodule of concern
7. Any illness or factor that will inhibit compliance with study participation

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with newly identified, solid lung nodule determined to be low-moderate risk of cancer.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Lung Nodule Diagnosis | Up to 24 months
  Malignant diagnosis through histology/pathology or benign diagnosis through histology/pathology, radiologic stability or radiologic confirmation of nodule resolution

CONTACTS AND LOCATIONS:
Overall Officials: Steven Springmeyer, Principal Investigator — Biodesix, Inc.; Gerard Silvestri, MD, Principal Investigator — Medical University of South Carolina
Locations (25):
- United States (23):
  - University of Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Connecticut
  - Beth Israel Deaconess, Boston, Connecticut
  - MedStar, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - The Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Washington University, St Louis, Missouri
  - Mount Sinai Health System, New York, New York
  - Northwell Health, New York, New York
  - The University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Coulmbus, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health, Greenville, South Carolina
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - McGill University Health Centre, Montreal, Quebec